CLINICAL TRIAL: NCT07099807
Title: Carbohydrate Mouth Rinsing Enhances Prefrontal Cortex Oxygenation and Cognitive Performance, Reducing Perceived Exertion During High-Intensity Exercise
Brief Title: Carbohydrate Mouth Rinsing and Cognitive Response During Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHA University (Other)
Responsible Party: Principal Investigator, Park Seung-Bo, CHA Bundang Medical Center, CHA University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Parks0524
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Exercise Performance of Fit Athletes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Carbohydrate Mouth Rinse (Experimental)
  Interventions: Behavioral: Carbohydrate Mouth Rinse
- Placebo Mouth Rinse (Placebo Comparator)
  Interventions: Behavioral: Placebo Mouth Rinse
- Music Listening (Experimental)
  Interventions: Behavioral: Music Listening

INTERVENTIONS:
Behavioral: Carbohydrate Mouth Rinse — A 6.4% maltodextrin solution (64 g/L) was prepared using Nutricost Maltodextrin Powder. Participants performed five mouth rinses per trial, each using 25 mL of the solution for 10 seconds before expectorating. Each rinse was followed by a 30-second rest. Participants were instructed not to swallow the solution. Rinsing procedure was standardized across all sessions.
  Arms: Carbohydrate Mouth Rinse
Behavioral: Placebo Mouth Rinse — A placebo solution containing 0.05 g/L of non-caloric sucralose in distilled water was used to match sweetness and viscosity of the CHO-MR. Participants performed five rinses of 25 mL for 10 seconds each, spitting out the solution after each rinse. 30-second rest intervals followed each rinse. Swallowing was not allowed. Rinse frequency, volume, and duration were standardized.
  Arms: Placebo Mouth Rinse
Behavioral: Music Listening — Participants listened to high-tempo music (120 bpm) for 15 minutes before exercise using standardized earbuds. Music was selected from a public YouTube playlist titled "120 BPM Best Dance Music for Running and Working Out." Volume was calibrated at 65 dB (50% of max device volume). Auditory conditions were standardized across all participants.
  Arms: Music Listening

SUMMARY:
This study investigates whether rinsing the mouth with a carbohydrate solution can improve brain oxygenation and cognitive function during high-intensity exercise. Eleven trained cyclists participated in multiple exercise sessions under different mouth rinse conditions. Brain oxygenation, perceived exertion, and cognitive performance were measured. The goal is to understand if this simple technique can support both physical and mental performance during demanding exercise.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 and 30 years
* Engaged in regular cycling training (≥5 sessions per week, ~4 hours per day)
* No known cardiovascular, neurological, or metabolic diseases
* Provided written informed consent

Exclusion Criteria:

* Current use of medication affecting cardiovascular or cognitive function
* Recent musculoskeletal injuries that affect cycling ability
* Smoking or excessive alcohol consumption
* Refusal or inability to comply with study procedures

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2025-02-28 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-17 (Actual)

PRIMARY OUTCOMES:
Changes in prefrontal cortex oxygenation (ΔO2Hb) | Immediately post-intervention and post-time trial (within same day)

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Bo Park, Principal Investigator — CHA University
Locations (1):
- CHA University, Human Performance Lab, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No